CLINICAL TRIAL: NCT00386165
Title: A Phase Ib, Randomized, Double-Blind, Placebo Controlled Study to Determine the Safety, Tolerance, Pharmacokinetic and Pharmacodynamic Effects of Single Doses of Larazotide Acetate (AT-1001) in Celiac Disease Subjects.
Brief Title: Safety Study of Larazotide Acetate to Treat Celiac Disease.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: 9 Meters Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLIN1001-002
Record Dates: First submitted 2006-10-09; First posted 2006-10-11 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Celiac Disease
Keywords: larazotide acetate
MeSH Terms: conditions — Celiac Disease | interventions — larazotide acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Larazotide acetate (Experimental): Larazotide acetate capsules: 12 mg QD x 3 days
  Interventions: Drug: larazotide acetate
- Placebo (Placebo Comparator): Placebo capsules: QD x 3 days
  Interventions: Drug: larazotide acetate

INTERVENTIONS:
Drug: larazotide acetate — larazotide acetate 4 mg capsules
  Other Names: AT-1001; INN-202

SUMMARY:
To demonstrate the safety, pharmacokinetics and efficacy of larazotide acetate in patients with controlled celiac disease on a gluten-free diet following a gluten challenge.

DETAILED DESCRIPTION:
CLIN1001-002 was a Phase 1b, randomized, double-blind, placebo controlled study to determine the safety, tolerance, pharmacokinetic and pharmacodynamic effects of single doses of larazotide acetate in subjects with celiac disease subjects. Study subjects were randomized (2:1) to receive single oral doses of larazotide acetate 12 mg or matching placebo once daily for 3 days. Subjects received a single-blinded gluten challenge (5 mg amygluten) on Day 2. Intestinal permeability was measured each day following dosing. Intestinal permeability was measured by administration of an oral sucrose, lactulose and mannitol solution followed by a 6-hour urine collection. Serial blood samples were collected for pharmacokinetic determinations at baseline and 2 and 3 hours post dose; for zonulin determinations at baseline (prior to first dose) and 3 hours post dose; and for cytokine determination at baseline and 3 hours post dose (Days 2 and 3 only) and on Day 7. Sucrose, lactulose, mannitol, zonulin and larazotide acetate concentrations were determined by validated analytical methods.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have been diagnosed with celiac disease by biopsy for ≥ 6 months (attending physician confirmation will be accepted in lieu of a biopsy report).
* Subject must be on a gluten-free diet for at least the past 6 months.

Exclusion Criteria:

* Subject has Anti-Tissue Transglutaminase (tTG) > 10 EU as measured by serology
* Subject intermittently consumes clinically significant quantities of non-steroidal anti-inflammatory agents ("NSAIDs") and proton-pump inhibitors, within the last 3 days prior to the treatment visit.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2005-11-29 (Actual); Primary Completion 2006-01-26 (Actual); Study Completion 2006-01-26 (Actual)

PRIMARY OUTCOMES:
Demonstrate the safety and tolerance of single doses of larazotide acetate in patients with controlled celiac disease on a gluten-free diet. | AEs were monitored throughout the study. Clinical laboratory testing was performed at scheduled times throughout the study. ECGs were measured at baseline, 3 hours post-dose on all study days and at the follow-up visit.
  Safety assessments included scheduled monitoring of adverse events (AEs), vital sign measurements, 12-lead ECG measurements, physical examinations, and clinical laboratory testing (chemistry, hematology, and urinalysis).
Determine whether quantifiable concentrations of larazotide acetate are present in plasma following single oral doses and to characterize the pharmacokinetic behavior of larazotide acetate in celiac disease subjects that are gluten-free and in remission | erial blood samples were collected for pharmacokinetic determinations at baseline and 2 and 3 hours post dose.
  Pharmacokinetic samples were taken to determine whether quantifiable concentrations of larazotide acetate were present in plasma following single oral doses and to characterize the pharmacokinetic behavior of larazotide acetate in celiac disease subjects.
Evaluate the effects of single doses of larazotide acetate on intestinal permeability ratios and zonulin levels | Intestinal permeability was measured each day following dosing. A gluten challenge was administered on Day 2.
  Intestinal permeability was measured by administration of an oral sucrose, lactulose and mannitol solution followed by urine and serum collection to measure urinary lactulose and mannitol, and serum zonulin concentrations as biomarkers.

SECONDARY OUTCOMES:
Self-reported measures of GI discomfort | Once daily on dosing days
  GI discomfort was reported by marking an "X" on a 10 cm linear line. Other GI Symptoms were assessed by subjects answering three questions related to bowel function.
Patient Global Assessment of Disease Status | At discharge from the clinic
  Subjects chose one of seven ordinal levels in response to a question related to any change in their disease status since being admitted to the clinic

CONTACTS AND LOCATIONS:
Overall Officials: Blake Paterson, MD, Study Chair — Alba Therapeutics
Locations (1):
- Parexel, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Paterson BM, Lammers KM, Arrieta MC, Fasano A, Meddings JB. The safety, tolerance, pharmacokinetic and pharmacodynamic effects of single doses of AT-1001 in coeliac disease subjects: a proof of concept study. Aliment Pharmacol Ther. 2007 Sep 1;26(5):757-66. doi: 10.1111/j.1365-2036.2007.03413.x. PMID 17697209